CLINICAL TRIAL: NCT06768346
Title: A Phase II, Open Label, Multicentre, Randomised Controlled Trial Comparing Hyperthermia Plus Mitomycin To Mitomycin Alone In Patients With Intermediate Risk Non-Muscle Invasive Bladder Cancer
Brief Title: Hyperthermic Intra-Vesical Chemotherapy
Acronym: HIVECII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-2013-04
Record Dates: First submitted 2017-08-25; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitomycin (No Intervention): Patients will receive six consecutive weekly instillations of Mitomycin followed by surveillance
- Hyperthermia+Mitomycin (Experimental): Patients will receive 6 weekly instillations of hyperthermia plus Mitomycin (HIVEC) using the COMBAT system, followed by surveillance cystoscopy.
  Interventions: Device: Hyperthermia will be delivered in combination with each instillation using the Combat BRS system

INTERVENTIONS:
Device: Hyperthermia will be delivered in combination with each instillation using the Combat BRS system — The Combat BRS system is a temperature controlled fluid recirculation system for the delivery of hyperthermic intravesical chemotherapy. The chemotherapy fluid is circulated in a closed system and warmed by an external isolated dry system using a novel innovative laminated aluminium foil heat exchanger with a small priming volume.
  Arms: Hyperthermia+Mitomycin

SUMMARY:
The purpose of the HIVEC II trial is to find out if the combination of the new technology called hyperthermia (the use of heat) and a drug called mitomycin is more effective than mitomycin alone which is the standard treatment for bladder cancer in reducing the chances of bladder cancer returning.

DETAILED DESCRIPTION:
The concept of hyperthermia plus MM has been demonstrated and a phase II randomized controlled trial of ablative HM versus MM using an alternative device (Synergo) has reported tumor ablation complete response (CR) rates in 66 % of tumors treated with hyperthermia plus mitomycin compared to 22% CR for MM mono-therapy.

Registered patients will be randomised to receive either Hyperthermia and Mitomycin or Mitomycin alone. Following treatment, patients will be followed up by surveillance cystoscopy for 24 months for disease recurrence. In the first year, the follow up visits will be every 3 months from the date of start of treatment and in the second year, the visits will be every 6 months.

The study also includes translational components to determine biomarkers of response to Heated Mitomycin. Urine samples will be collected prior to surveillance cystoscopies.

This study will address the problem of how to improve the disease free survival in patients with intermediate-risk NMIBC, the treatment must have acceptable side-effects, low toxicity, and show a significant benefit over MM alone.

ELIGIBILITY:
Inclusion Criteria:

1. New or Recurrence of intermediate risk NMIBC following TURBT defined as;

   * Grade 2 or grade 1 stage Ta or T1 disease*.
   * Any grade G2 or G1 other than Low risk
2. Age ≥ 18 yrs
3. WHO performance status 0, 1, 2, 3
4. Pre-treatment haematology and biochemistry values within acceptable limits:

   * Haemoglobin > or =10 g/dL
   * Neutrophil count > or =1.5 x 109/L
   * Platelets > or = 100 x 109/L
   * WBC > or = 3.0 x 109/L or ANC > or = 1.5 x 109/L
   * Serum creatinine < 1.5 x UNL
5. Negative pregnancy test for women of child-bearing potential.
6. Available for long-term follow-up.
7. Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
8. Written informed consent.

Exclusion Criteria:

1. Grade 3 TCC
2. Carcinoma in situ.
3. New solitary Ta G1 (small)
4. New solitary Ta G2 (small)
5. Previous intravesical chemotherapy in the past 6 months, other than single instillation post-TUR.
6. Bladder capacity <200cc.
7. UCC involving the prostatic urethra or upper urinary tract.
8. > or =T2 UCC
9. Known allergy to mitomycin
10. Pregnant or lactating women or women of childbearing potential unwilling or unable to use adequate non-hormonal contraception.
11. Other malignancy within the past five years, except: non-melanomatous skin cancer cured by excision, adequately treated carcinoma in situ of the cervix or DCIS/LCIS of the breast or prostate cancer with more than 5yrs life expectancy or any non lifethreatening tumours that have been curatively treated.
12. Concurrent chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2014-05-08 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
To determine if HIVEC increases disease-free survival at 24 months compared to the comparator arm of MM alone. | After the last patient has completed 24 months follow-up
  The interval in whole days between the date of randomisation into the trial and the earliest of date of detection of recurrent disease, or date (known as Disease- free survival) will be measured.
  of death from any cause.

SECONDARY OUTCOMES:
To determine if HIVEC reduces the risk of recurrence at 3 months compared to the control arm, for patients with intermediate risk disease. | At the end of study - After all patients have been followed-up for at least 2 years
  The recurrence of tumor at 3 months will be calculated as a time to event outcome. recurrence of tumor at 3 months can predict subsequent recurrence and as a surrogate outcome will be monitored as a secondary measure.
Progression Free Survival | At the end of study - After all patients have been followed-up for at least 2 years
  Progression-free survival: Defined as the interval in whole days between the date of randomisation into the trial and the earliest of date of detection of disease progression, or date of death from any cause
Recurrence-free survival. | At the end of study - After all patients have been followed-up for at least 2 years
  Recurrence free survival will be measured in patients with papillary disease only. It is defined in the same way as disease free survival, with the important distinction that CIS at the first three-month post-treatment will not be included as an event, but rather considered a treatment failure and will be censored.
To determine if Heated Mytomycin reduces the risk of progression to invasive disease compared to the control arm. | After all patients have been followed-up for at least 2 years
  Progression Free Survival will be compared between the 2 arms. Progression free survival is defined as the interval in whole days between the date of randomisation into the trial and the earliest of date of detection of disease progression, or date of death from any cause.
To compare overall and disease-specific survival between the Heated Mytomycin and the control arm. | At the end of study - After all patients have been followed-up for at least 2 years
  Overall and Disease specific survival will be measured in terms of time interval. Overall survival: Defined as the interval in whole days between the date of randomisation into the trial and date of death from any cause; patients who do not die during the course of the trial will be censored at the last follow-up date. Disease specific survival: Defined as the interval in whole days between the date of randomisation into the trial and date of death due to bladder cancer. Patients who do not die during the course of the trial will be censored at the last follow-up date. Patients who die of other causes will be censored at date of death due to other cause.
To define the safety and tolerability of Heated Mytomycin in this patient population. | At the end of study - After all patients have been followed-up for at least 2 years
  Safety and Tolerability will be reported through the number of adverse events. This will include assessment of frequency, severity and nature of adverse events and the treatment received
To compare QOL between the Heated Mytomycin and the control arms. | After all patients have been followed-up for at least 2 years
  Quality of life will be assessed at study entry and every three months using the questionnaires. The questionnaires collects information about side effects and symptoms as well as measures of function and overall well being. For each part, a set scale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Dr John Kelly, Principal Investigator — Queen Mary University of London
Locations (14):
- United Kingdom (14):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Western General Hospital, Edinburgh, Edinburgh
  - Royal Surrey County Hospital NHS Foudation Trust, Guildford
  - The Clatterbridge Cancer Centre, Liverpool
  - Barnet Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - University College London Hospital, London., London
  - University Hospital of South Manchester, Manchester
  - South Tees NHS Trust - James Cook University Hospital, Middlesbrough
  - Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich
  - Derriford Hospital, Plymouth
  - Portsmouth Hospitals NHS Trust - Queen Alexandra Hospital, Portsmouth
  - East Surrey Hospital, Redhill
  - New Cross Hospital, Wolverhampton

REFERENCES:
- See also: Related Info — https://www.isrctn.com/ISRCTN23639415